CLINICAL TRIAL: NCT05262751
Title: A Phase I Study for Formulation Selection and Subsequent Optimization of Two Different Oral Formulations of Nintedanib in Healthy Male Subjects (Open-label, Randomised, Single-dose Study in Three Parts)
Brief Title: A Study in Healthy Men to Find the Best Formulation for Once Daily Intake of Nintedanib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1199-0452; 2021-003152-16 (EudraCT Number)
Record Dates: First submitted 2022-03-01; First posted 2022-03-02 (Actual); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Healthy
MeSH Terms: interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Each participant received: Nintedanib formulation 1: Monolithic Nintedanib Modified Release Tablet (MR1) as two Prototypes (MR1-1 and MR1-2), compared to the reference (R) treatment: Nintedanib formulation 3: Ofev®.
  Interventions: Drug: Ofev®; Drug: Nintedanib formulation 1
- Cohort 2 (Experimental): Nintedanib formulation 2: Polyox Nintedanib Modified Release Tablet (MR2) as two Prototypes (MR2-1 and MR2-2) compared to the reference (R) treatment: Nintedanib formulation 3: Ofev®.
  Interventions: Drug: Ofev®; Drug: Nintedanib formulation 2

INTERVENTIONS:
Drug: Ofev® — Ofev®
  Other Names: Nintedanib
Drug: Nintedanib formulation 1 — Nintedanib formulation 1: Monolithic Nintedanib Modified Release Tablet (MR1) as two Prototypes (MR1-1 and MR1-2).
  Arms: Cohort 1
Drug: Nintedanib formulation 2 — Nintedanib formulation 2: Polyox Nintedanib Modified Release Tablet (MR2) as two Prototypes (MR2-1 and MR2-2).
  Arms: Cohort 2

SUMMARY:
The main objective of this trial is to assess single dose drug exposure of several newly developed formulation prototypes of Nintedanib compared to Ofev® following oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects (Caucasian and Black only) according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiograms (ECG) and clinical laboratory tests.
* Age of 18 to 55 years (inclusive).
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive) and absolute body weight of at least 65 kg.
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation.
* Non-smokers for at least 6 months.
* Subjects who are sexually active must use with their partner, highly effective contraception from the time of administration of trial medication until 30 days after administration of trial medication. Adequate methods are:

  * Condoms plus use of hormonal contraception by the female partner that started at least 2 months prior to administration of trial medication (e.g., implants, injectables, combined oral or vaginal contraceptives, intrauterine device) or;
  * Condoms plus surgical sterilization (vasectomy at least 1 year prior to enrolment) or;
  * Condoms plus surgically sterilised partner (including hysterectomy) or;
  * Condoms plus intrauterine device or;
  * Condoms plus partner of non-childbearing potential (including homosexual men). Subjects are required to use condoms to prevent unintended exposure of the partner (both, male and female) to the study drug via seminal fluid. Male subjects should use a condom throughout the study and for 30 days after last Investigational Medicinal Product (IMP) administration. Alternatively, true abstinence is acceptable when it is in line with the subject's preferred and usual lifestyle. If a subject is usually not sexually active but becomes active with their partner, they must comply with the contraceptive requirements detailed above.

Male subjects should not donate sperm for the duration of the study and for at least 30 days after last IMP administration. Male subjects with pregnant or lactating partners are allowed.

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator.
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm).
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance.
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results.
* Liver enzymes (Aspartate amino transferase (AST) and Alanine amino transferase (ALT)) above upper limit of normal at the screening examination.
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator.
* Clinically significant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, dermatological or hormonal disorders. Subjects with Gilbert's syndrome are not permitted.
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair).

Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was a randomised, open-label, crossover, single-dose (once daily [qd] for test and twice daily [bid] for reference treatment) study in up to 3 parts; trial part 1: 2 parallel groups (Cohort 1, Cohort 2), each a randomised three-period crossover; trial part 2 (optional): one group of randomised three-period crossover; trial part 3 (optional): one group of randomised two-period crossover. Parts 2 and 3 were not performed. The trial was stopped as per protocol during trial part 1.
Pre-assignment Details: Only participants that met all the study inclusion and none of the exclusion criteria were to be entered in the study. All participants were free to withdraw from the clinical trial at any time for any reason given. Close monitoring of all participants was adhered to throughout the trial conduct. Rescue medication was allowed for all participants as required.
Groups:
- Cohort 1: R | MR1-1 | MR1-2: In this arm participants were treated at 3 treatment visits (= 3 treatment periods). There was a washout period of at least 14 days between each treatment visit, i.e. the morning dose in the preceding treatment period and the morning dose in the following treatment period were separated by at least 14 days.
  Treatments:
  * First: R, a low oral dose of Ofev® capsule bid with 240 milliliter (ml) of water after a light breakfast and dinner, respectively;
  * Second: MR1-1, a single medium oral dose of Nintedanib MR1-1 tablet with 240 ml water in the morning after a light breakfast;
  * Third: MR1-2, a single medium oral dose of Nintedanib MR1-2 tablet with 240 ml water in the morning after a light breakfast.
  Abbreviations:
  R=Reference=Ofev® capsules, MR1-1=Monolithic Nintedanib Modified Release Prototype 1 Tablet, MR1-2=Monolithic Nintedanib Modified Release Prototype 2 Tablet.
- Cohort 1: MR1-2 | R | MR1-1: In this arm participants were treated at 3 treatment visits (= 3 treatment periods). There was a washout period of at least 14 days between each treatment visit, i.e. the morning dose in the preceding treatment period and the morning dose in the following treatment period were separated by at least 14 days.
  Treatments:
  * First: MR1-2, a single medium oral dose of Nintedanib MR1-2 tablet with 240 ml water in the morning after a light breakfast;
  * Second: R, a low oral dose of Ofev® capsule bid with 240 ml of water after a light breakfast and dinner, respectively;
  * Third: MR1-1, a single medium oral dose of Nintedanib MR1-1 tablet with 240 ml water in the morning after a light breakfast.
- Cohort 1: MR1-1 | MR1-2 | R: In this arm participants were treated at 3 treatment visits (= 3 treatment periods). There was a washout period of at least 14 days between each treatment visit, i.e. the morning dose in the preceding treatment period and the morning dose in the following treatment period were separated by at least 14 days.
  Treatments:
  * First: MR1-1, a single medium oral dose of Nintedanib MR1-1 tablet with 240 ml water in the morning after a light breakfast;
  * Second: MR1-2, a single medium oral dose of Nintedanib MR1-2 tablet with 240 ml water in the morning after a light breakfast;
  * Third: R, a low oral dose of Ofev® capsule bid with 240 ml of water after a light breakfast and dinner, respectively.
- Cohort 2: R | MR2-1 | MR2-2: In this arm participants were treated at 3 treatment visits (= 3 treatment periods). There was a washout period of at least 14 days between each treatment visit, i.e. the morning dose in the preceding treatment period and the morning dose in the following treatment period were separated by at least 14 days.
  Treatments:
  * First: R, a low oral dose of Ofev® capsule bid with 240 ml of water after a light breakfast and dinner, respectively;
  * Second: MR2-1, a single medium oral dose of Nintedanib MR2-1 tablet with 240 ml water in the morning after a light breakfast;
  * Third: MR2-2, a single medium oral dose of Nintedanib MR2-2 tablet with 240 ml water in the morning after a light breakfast.
  Abbreviations:
  R=Reference=Ofev® capsules, MR2-1=Polyox Nintedanib Modified Release Prototype 1 Tablet, MR2-2=Polyox Nintedanib Modified Release Prototype 2 Tablet.
- Cohort 2: MR2-2 | R | MR2-1: In this arm participants were treated at 3 treatment visits (= 3 treatment periods). There was a washout period of at least 14 days between each treatment visit, i.e. the morning dose in the preceding treatment period and the morning dose in the following treatment period were separated by at least 14 days.
  Treatments:
  * First: MR2-2, a single medium oral dose of Nintedanib MR2-2 tablet with 240 ml water in the morning after a light breakfast;
  * Second: R, a low oral dose of Ofev® capsule bid with 240 ml of water after a light breakfast and dinner, respectively;
  * Third: MR2-1, a single medium oral dose of Nintedanib MR2-1 tablet with 240 ml water in the morning after a light breakfast.
- Cohort 2: MR2-1 | MR2-2 | R: In this arm participants were treated at 3 treatment visits (= 3 treatment periods). There was a washout period of at least 14 days between each treatment visit, i.e. the morning dose in the preceding treatment period and the morning dose in the following treatment period were separated by at least 14 days.
  Treatments:
  * First: MR2-1, a single medium oral dose of Nintedanib MR2-1 tablet with 240 ml water in the morning after a light breakfast;
  * Second: MR2-2, a single medium oral dose of Nintedanib MR2-2 tablet with 240 ml water in the morning after a light breakfast;
  * Third: R, a low oral dose of Ofev® capsule bid with 240 ml of water after a light breakfast and dinner, respectively.
Period: Treatment Period 1
Arm/Group | Cohort 1: R | MR1-1 | MR1-2 | Cohort 1: MR1-2 | R | MR1-1 | Cohort 1: MR1-1 | MR1-2 | R | Cohort 2: R | MR2-1 | MR2-2 | Cohort 2: MR2-2 | R | MR2-1 | Cohort 2: MR2-1 | MR2-2 | R
Started | 3 | 2 | 2 | 5 | 5 | 4
Completed | 3 | 2 | 2 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | Cohort 1: R | MR1-1 | MR1-2 | Cohort 1: MR1-2 | R | MR1-1 | Cohort 1: MR1-1 | MR1-2 | R | Cohort 2: R | MR2-1 | MR2-2 | Cohort 2: MR2-2 | R | MR2-1 | Cohort 2: MR2-1 | MR2-2 | R
Started | 3 | 2 | 2 | 5 | 5 | 4
Completed | 3 | 2 | 2 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Cohort 1: R | MR1-1 | MR1-2 | Cohort 1: MR1-2 | R | MR1-1 | Cohort 1: MR1-1 | MR1-2 | R | Cohort 2: R | MR2-1 | MR2-2 | Cohort 2: MR2-2 | R | MR2-1 | Cohort 2: MR2-1 | MR2-2 | R
Started | 3 | 2 | 2 | 5 | 5 | 4
Completed | 3 | 2 | 2 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | Cohort 1: R | MR1-1 | MR1-2 | Cohort 1: MR1-2 | R | MR1-1 | Cohort 1: MR1-1 | MR1-2 | R | Cohort 2: R | MR2-1 | MR2-2 | Cohort 2: MR2-2 | R | MR2-1 | Cohort 2: MR2-1 | MR2-2 | R
Started | 3 | 2 | 2 | 5 | 5 | 4
Completed | 2 | 2 | 2 | 5 | 5 | 4
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Cohort 1: R | MR1-1 | MR1-2 | Cohort 1: MR1-2 | R | MR1-1 | Cohort 1: MR1-1 | MR1-2 | R | Cohort 2: R | MR2-1 | MR2-2 | Cohort 2: MR2-2 | R | MR2-1 | Cohort 2: MR2-1 | MR2-2 | R
Started | 2 | 2 | 2 | 5 | 5 | 4
Treated | 2 | 1 | 2 | 5 | 5 | 4
Completed | 2 | 1 | 2 | 5 | 5 | 4
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Not treated because of an adverse event | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all participants who were randomized and treated with at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: R | MR1-1 | MR1-2 | Cohort 1: MR1-2 | R | MR1-1 | Cohort 1: MR1-1 | MR1-2 | R | Cohort 2: R | MR2-1 | MR2-2 | Cohort 2: MR2-2 | R | MR2-1 | Cohort 2: MR2-1 | MR2-2 | R | Total
Number analyzed (Participants) | 3 | 2 | 2 | 5 | 5 | 4 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.7 (16.2) | 36.5 (20.5) | 44.5 (7.8) | 35.8 (8.6) | 32.2 (9.2) | 34.5 (11.6) | 36.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 2 | 2 | 5 | 5 | 4 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 2 | 5 | 5 | 4 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 3 | 2 | 1 | 5 | 4 | 4 | 19
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of 3 Different Formulations of Nintedanib (MR1, MR2 and Ofev®) in Plasma Over the Time Interval From 0 Extrapolated to Infinity Which Includes Also the Second Nintedanib (Ofev®) Dose of the Day (AUC₀-∞)
Description: The area under the concentration-time curve over the time interval from 0 [first dose] extrapolated to infinity (AUC₀-∞) was analyzed in 3 different formulations of Nintedanib (MR1, MR2 and Ofev®) and in two cohorts:
  * Cohort 1: Nintedanib formulation 1: Monolithic Nintedanib Modified Release Tablet (MR1) as two Prototypes (MR1-1 and MR1-2),
  * Cohort 2: Nintedanib formulation 2: Polyox Nintedanib Modified Release Tablet (MR2) as two Prototypes (MR2-1 and MR2-2), and each compared to the reference (R) treatment: Nintedanib formulation 3: Ofev® capsules.
  The adjusted geometric least squares mean and adjusted geometric standard error were calculated by an analysis of variance (ANOVA) model on the logarithmic scale.
Time Frame: Within 3 hours (h) prior and 1, 2, 3, 4, 6, 8, 10, 12, 13 (except MR1, MR2), 14, 15, 16, 17 (except R), 18, 20, 22, 24, 34, 48, 58, and 72 h after administration.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This set includes all subjects in the treated set (TS) who provide at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Only subjects with available PK data were included in this analysis.
Measure: Geometric Least Squares Mean (Standard Error); unit: Hours times nanogram per milliliter
Groups:
- Cohort 1: Reference (R): A low oral dose of Ofev® (Reference (R)) capsule bid was administered with 240 millilitre (ml) of water after a light breakfast and dinner, respectively on one day.
- Cohort 1: Test Treatment 1 (MR1-1): A single medium oral dose of Monolithic Nintedanib Modified Release Prototype 1 Tablet (MR1-1) was administered with 240 ml water in the morning after a light breakfast on one day.
- Cohort 1: Test Treatment 2 (MR1-2): A single medium oral dose of Monolithic Nintedanib Modified Release Prototype 2 Tablet (MR1-2) was administered with 240 ml water in the morning after a light breakfast on one day.
- Cohort 2: Reference (R): A low oral dose of Ofev® capsule (R) bid was administered with 240 ml of water after a light breakfast and dinner, respectively on one day.
- Cohort 2: Test Treatment 1 (MR2-1): A single medium oral dose of Polyox Nintedanib Modified Release Prototype 1 Tablet (MR2-1) was administered with 240 ml water in the morning after a light breakfast on one day.
- Cohort 2: Test Treatment 2 (MR2-2): A single medium oral dose of Nintedanib Polyox Nintedanib Modified Release Prototype 2 Tablet (MR2-2) was administered with 240 ml water in the morning after a light breakfast on one day.
Arm/Group | Cohort 1: Reference (R) | Cohort 1: Test Treatment 1 (MR1-1) | Cohort 1: Test Treatment 2 (MR1-2) | Cohort 2: Reference (R) | Cohort 2: Test Treatment 1 (MR2-1) | Cohort 2: Test Treatment 2 (MR2-2)
Number analyzed (Participants) | 7 | 3 | 4 | 13 | 12 | 11
Hours times nanogram per milliliter | 359.80 (NA) — Adjusted geometric standard error = 1.18 | 60.04 (NA) — Adjusted geometric standard error = 1.46 | 48.72 (NA) — Adjusted geometric standard error = 1.26 | 241.32 (NA) — Adjusted geometric standard error = 1.15 | 100.88 (NA) — Adjusted geometric standard error = 1.16 | 103.55 (NA) — Adjusted geometric standard error = 1.16
Statistical Analysis 1: Comparison: Cohort 1: Reference (R) vs Cohort 1: Test Treatment 1 (MR1-1); Analysis of Variance (ANOVA) model (logarithmic scale) with the effects: sequence, subjects within sequences, period, and treatment. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; Test type: Other; gMean Ratio = 16.69, 90% CI 2-sided [7.28 to 38.24] — gMean Ratio: MR1-1/R. Intra-individual Geometric coefficient of variation [%] = 34.1
Statistical Analysis 2: Comparison: Cohort 1: Reference (R) vs Cohort 1: Test Treatment 2 (MR1-2); [analysis description as in outcome 1, analysis 1]; Test type: Other; gMean Ratio = 13.54, 90% CI 2-sided [8.10 to 22.64] — gMean Ratio: MR1-2/R. Intra-individual Geometric coefficient of variation [%] = 34.1
Statistical Analysis 3: Comparison: Cohort 2: Reference (R) vs Cohort 2: Test Treatment 1 (MR2-1); [analysis description as in outcome 1, analysis 1]; Test type: Other; gMean Ratio = 41.80, 90% CI 2-sided [34.24 to 51.04] — gMean Ratio: MR2-1/R. Intra-individual Geometric coefficient of variation [%] = 28.4
Statistical Analysis 4: Comparison: Cohort 2: Reference (R) vs Cohort 2: Test Treatment 2 (MR2-2); [analysis description as in outcome 1, analysis 1]; Test type: Other; gMean Ratio = 42.91, 90% CI 2-sided [34.90 to 52.76] — gMean Ratio: MR2-2/R. Intra-individual Geometric coefficient of variation [%] = 28.4

2. Secondary Outcome: Area Under the Concentration-time Curve of 3 Different Formulations of Nintedanib (MR1, MR2 and Ofev®) in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC₀-tz)
Description: The area under the concentration-time curve over the time interval from 0 to the last quantifiable data point (AUC₀-tz) was analyzed in 3 different formulations of Nintedanib (MR1, MR2 and Ofev®) and in two cohorts:
  * Cohort 1: Nintedanib formulation 1: Monolithic Nintedanib Modified Release Tablet (MR1) as two Prototypes (MR1-1 and MR1-2),
  * Cohort 2: Nintedanib formulation 2: Polyox Nintedanib Modified Release Tablet (MR2) as two Prototypes (MR2-1 and MR2-2), and each compared to the reference (R) treatment: Nintedanib formulation 3: Ofev® capsules.
  The adjusted geometric least squares mean and adjusted geometric standard error were calculated by an analysis of variance (ANOVA) model on the logarithmic scale.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: Hours times nanogram per milliliter
Arm/Group | Cohort 1: Reference (R) | Cohort 1: Test Treatment 1 (MR1-1) | Cohort 1: Test Treatment 2 (MR1-2) | Cohort 2: Reference (R) | Cohort 2: Test Treatment 1 (MR2-1) | Cohort 2: Test Treatment 2 (MR2-2)
Number analyzed (Participants) | 7 | 6 | 6 | 13 | 14 | 14
Hours times nanogram per milliliter | 326.48 (NA) — Adjusted geometric standard error = 1.21 | 30.54 (NA) — Adjusted geometric standard error = 1.24 | 40.51 (NA) — Adjusted geometric standard error = 1.23 | 226.69 (NA) — Adjusted geometric standard error = 1.19 | 85.91 (NA) — Adjusted geometric standard error = 1.19 | 81.35 (NA) — Adjusted geometric standard error = 1.19
Statistical Analysis 1: Comparison: Cohort 1: Reference (R) vs Cohort 1: Test Treatment 1 (MR1-1); [analysis description as in outcome 1, analysis 1]; Test type: Other; gMean Ratio = 9.36, 90% CI 2-sided [5.91 to 14.80] — gMean Ratio: MR1-1/R. Intra-individual Geometric coefficient of variation [%] = 44.8
Statistical Analysis 2: Comparison: Cohort 1: Reference (R) vs Cohort 1: Test Treatment 2 (MR1-2); [analysis description as in outcome 1, analysis 1]; Test type: Other; gMean Ratio = 12.41, 90% CI 2-sided [7.93 to 19.43] — gMean Ratio: MR1-2/R. Intra-individual Geometric coefficient of variation [%] = 44.8
Statistical Analysis 3: Comparison: Cohort 2: Reference (R) vs Cohort 2: Test Treatment 1 (MR2-1); [analysis description as in outcome 1, analysis 1]; Test type: Other; gMean Ratio = 37.90, 90% CI 2-sided [29.25 to 49.11] — gMean Ratio: MR2-1/R. Intra-individual Geometric coefficient of variation [%] = 40.4
Statistical Analysis 4: Comparison: Cohort 2: Reference (R) vs Cohort 2: Test Treatment 2 (MR2-2); [analysis description as in outcome 1, analysis 1]; Test type: Other; gMean Ratio = 35.89, 90% CI 2-sided [27.66 to 46.55] — gMean ratio: MR2-2/R. Intra-individual Geometric coefficient of variation [%] = 40.4

3. Secondary Outcome: Maximum Measured Concentration of 3 Different Formulations of Nintedanib (MR1, MR2 and Ofev®) in Plasma Within the 24h Dosing Interval (Cmax)
Description: The maximum measured concentration in plasma was analyzed in 3 different formulations of Nintedanib (MR1, MR2 and Ofev®) and in two cohorts:
  * Cohort 1: Nintedanib formulation 1: Monolithic Nintedanib Modified Release Tablet (MR1) as two Prototypes (MR1-1 and MR1-2),
  * Cohort 2: Nintedanib formulation 2: Polyox Nintedanib Modified Release Tablet (MR2) as two Prototypes (MR2-1 and MR2-2), and each compared to the reference (R) treatment: Nintedanib formulation 3: Ofev® capsules.
  The adjusted geometric least squares mean and adjusted geometric standard error were calculated by an analysis of variance (ANOVA) model on the logarithmic scale.
Time Frame: Within 3 hours (h) prior and 1.0, 2.0, 3.0, 4.0, 6.0, 8.0, 10.0, 12.0, 13.0 (except MR1, MR2), 14.0, 15.0, 16.0, 17.0 (except R), 18.0, 20.0, 22.0, 24.0, 34.0, 48.0, 58.0, and 72 h after administration
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: Nanogram per milliliter
Groups:
- Cohort 2: Test Treatment 2 (MR2-2): A single medium oral dose of Polyox Nintedanib Modified Release Prototype 1 Tablet (MR2-1) was administered with 240 ml water in the morning after a light breakfast on one day.
Arm/Group | Cohort 1: Reference (R) | Cohort 1: Test Treatment 1 (MR1-1) | Cohort 1: Test Treatment 2 (MR1-2) | Cohort 2: Reference (R) | Cohort 2: Test Treatment 1 (MR2-1) | Cohort 2: Test Treatment 2 (MR2-2)
Number analyzed (Participants) | 7 | 6 | 6 | 13 | 14 | 14
Nanogram per milliliter | 32.02 (NA) — Adjusted geometric standard error = 1.32 | 3.87 (NA) — Adjusted geometric standard error = 1.35 | 7.66 (NA) — Adjusted geometric standard error = 1.34 | 17.55 (NA) — Adjusted geometric standard error = 1.19 | 12.03 (NA) — Adjusted geometric standard error = 1.18 | 11.73 (NA) — Adjusted geometric standard error = 1.18
Statistical Analysis 1: Comparison: Cohort 1: Reference (R) vs Cohort 1: Test Treatment 1 (MR1-1); [analysis description as in outcome 1, analysis 1]; Test type: Other; gMean Ratio = 12.09, 90% CI 2-sided [6.73 to 21.71] — gMean Ratio: MR1-1/R. Intra-individual Geometric coefficient of variation [%] = 58.8
Statistical Analysis 2: Comparison: Cohort 1: Reference (R) vs Cohort 1: Test Treatment 2 (MR1-2); [analysis description as in outcome 1, analysis 1]; Test type: Other; gMean Ratio = 23.94, 90% CI 2-sided [13.51 to 42.42] — gMean Ratio: MR1-2/R. Intra-individual Geometric coefficient of variation [%] = 58.8
Statistical Analysis 3: Comparison: Cohort 2: Reference (R) vs Cohort 2: Test Treatment 1 (MR2-1); [analysis description as in outcome 1, analysis 1]; Test type: Other; gMean Ratio = 68.55, 90% CI 2-sided [50.07 to 93.86] — gMean ratio: MR2-1/R. Intra-individual Geometric coefficient of variation [%] = 50.0
Statistical Analysis 4: Comparison: Cohort 2: Reference (R) vs Cohort 2: Test Treatment 2 (MR2-2); [analysis description as in outcome 1, analysis 1]; Test type: Other; gMean Ratio = 66.85, 90% CI 2-sided [48.77 to 91.64] — gMean ratio: MR2-2/R. Intra-individual Geometric coefficient of variation [%] = 50.0

4. Secondary Outcome: Concentration of 3 Different Formulations of Nintedanib (MR1, MR2 and Ofev®) in Plasma 24 Hours After the First Dose (C₂₄)
Description: The measured concentration in plasma 24 hours after first administration was analyzed in 3 different formulations of Nintedanib (MR1, MR2 and Ofev®) and in two cohorts:
  * Cohort 1: Nintedanib formulation 1: Monolithic Nintedanib Modified Release Tablet (MR1) as two Prototypes (MR1-1 and MR1-2),
  * Cohort 2: Nintedanib formulation 2: Polyox Nintedanib Modified Release Tablet (MR2) as two Prototypes (MR2-1 and MR2-2), and each compared to the reference (R) treatment: Nintedanib formulation 3: Ofev® capsules.
  The adjusted geometric least squares mean and adjusted geometric standard error were calculated by an analysis of variance (ANOVA) model on the logarithmic scale.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: Nanogram per milliliter
Arm/Group | Cohort 1: Reference (R) | Cohort 1: Test Treatment 1 (MR1-1) | Cohort 1: Test Treatment 2 (MR1-2) | Cohort 2: Reference (R) | Cohort 2: Test Treatment 1 (MR2-1) | Cohort 2: Test Treatment 2 (MR2-2)
Number analyzed (Participants) | 7 | 5 | 5 | 13 | 13 | 12
Nanogram per milliliter | 5.48 (NA) — Adjusted geometric standard error = 1.15 | 0.66 (NA) — Adjusted geometric standard error = 1.18 | 0.77 (NA) — Adjusted geometric standard error = 1.17 | 4.10 (NA) — Adjusted geometric standard error = 1.14 | 1.32 (NA) — Adjusted geometric standard error = 1.14 | 1.29 (NA) — Adjusted geometric standard error = 1.14
Statistical Analysis 1: Comparison: Cohort 1: Reference (R) vs Cohort 1: Test Treatment 1 (MR1-1); [analysis description as in outcome 1, analysis 1]; Test type: Other; gMean Ratio = 11.96, 90% CI 2-sided [8.88 to 16.11] — gMean ratio: MR1-1/R. Intra-individual Geometric coefficient of variation [%] = 23.5
Statistical Analysis 2: Comparison: Cohort 1: Reference (R) vs Cohort 1: Test Treatment 2 (MR1-2); [analysis description as in outcome 1, analysis 1]; Test type: Other; gMean Ratio = 13.98, 90% CI 2-sided [10.59 to 18.46] — gMean ratio: MR1-2/R. Intra-individual Geometric coefficient of variation [%] = 23.5
Statistical Analysis 3: Comparison: Cohort 2: Reference (R) vs Cohort 2: Test Treatment 1 (MR2-1); [analysis description as in outcome 1, analysis 1]; Test type: Other; gMean Ratio = 32.13, 90% CI 2-sided [26.46 to 39.01] — gMean ratio: MR2-1/R. Intra-individual Geometric coefficient of variation [%] = 29.3
Statistical Analysis 4: Comparison: Cohort 2: Reference (R) vs Cohort 2: Test Treatment 2 (MR2-2); [analysis description as in outcome 1, analysis 1]; Test type: Other; gMean Ratio = 31.38, 90% CI 2-sided [25.71 to 38.30] — gMean ratio: MR2-2/R. Intra-individual Geometric coefficient of variation [%] = 29.3

ADVERSE EVENTS:
Time Frame: From first drug administration in this period to at least 14 days thereafter OR until next drug administration of the following period, whatever occurred first, up to 22 days after last drug administration.
Description: Treated set (TS): The treated set included all participants who were randomized and treated with at least one dose of study drug.
Arm/Group | Cohort 1: Reference (R) | Cohort 1: Test Treatment 1 (MR1-1) | Cohort 1: Test Treatment 2 (MR1-2) | Cohort 2: Reference (R) | Cohort 2: Test Treatment 1 (MR2-1) | Cohort 2: Test Treatment 2 (MR2-2)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 3/7 | 1/6 | 0/6 | 4/14 | 4/14 | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Reference (R) (N=7) | Cohort 1: Test Treatment 1 (MR1-1) (N=6) | Cohort 1: Test Treatment 2 (MR1-2) (N=6) | Cohort 2: Reference (R) (N=14) | Cohort 2: Test Treatment 1 (MR2-1) (N=14) | Cohort 2: Test Treatment 2 (MR2-2) (N=14)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 2 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
As per protocol Parts 2 and 3 were not performed. The trial was stopped as per protocol during trial Part 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT05262751/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT05262751/SAP_001.pdf